CLINICAL TRIAL: NCT01123356
Title: Phase 2 Trial of Intracycle Sequential Ofatumumab and Lenalidomide for the Treatment of Chronic Lymphocytic Leukemia in Patients Previously Exposed to Rituximab
Brief Title: Treatment of Chronic Lymphocytic Leukemia in Patients Previously Exposed to Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: GlaxoSmithKline (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101376 OFT113297
Record Dates: First submitted 2010-05-04; First posted 2010-05-14 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Relapsed chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oratumumab and Lenalidomide (Experimental): Single arm, non randomized study
  Ofatumumab, Lenalidomide: -Ofatumumab 2000 mg (300 mg on first cycle) IV on day 1.
  * Lenalidomide 10 mg (5 mg on first cycle) PO days 8-28.
  * Treatment to be administered for up to 6 cycles
  Interventions: Drug: Ofatumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ofatumumab — * Ofatumumab 2000 mg (300 mg on first cycle) IV on day 1 for up to 6 cycles (28 day cycles)
  * Treatment to be administered for up to 6 cycles
  Other Names: Arzerra
Drug: Lenalidomide — -Lenalidomide 10 mg (5 mg on first cycle) PO days 8-28 for up to 6 cycles (28 day cycles)
  Other Names: Revlimid

SUMMARY:
The purpose of this research is to evaluate the safety and effectiveness of the drugs lenalidomide and ofatumumab in the treatment of chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have confirmed diagnosis of chronic lymphocytic leukemia (CLL).
2. Prior therapy with at least one regimen containing rituximab
3. Age > 18 years.
4. Life expectancy greater than 12 months.
5. ECOG performance status <2
6. Patients must have normal organ function as defined in the protocol.
7. Patients must have adequate bone marrow function as defined in the protocol.
8. Ability to understand and the willingness to sign a written informed consent document.
9. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
10. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks or received any monoclonal antibody within 6 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents or other anti-cancer agents or treatments.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ofatumumab or lenalidomide.
4. Uncontrolled concomitant illness.
5. Pregnant women are excluded from this study because lenalidomide is believed to be teratogenic.
6. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ofatumumab or lenalidomide.
7. Prior treatment with lenalidomide
8. Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome. Subjects may be enrolled upon correction of electrolyte abnormalities.
9. All patients will undergo screening for hepatitis B and may or may not be eligible based on the results as outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oratumumab and Lenalidomide
Started | 21
Completed | 14
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oratumumab and Lenalidomide
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Obtain early assessment of the efficacy of the intracycle sequential administration of ofatumumab and lenalidomide in the treatment of chronic lymphocytic leukemia (CLL) after prior use of rituximab. Response was categorized according to the IW-CLL criteria which includes the following: Complete remission (CR), CR with incomplete marrow recovery (CRi)Partial remission (PR), Progressive disease (PD), Stable disease (SD).
  Overall response rate was defined as those who experienced a response of CR, CRi or PR.
Time Frame: 30 Weeks
Population: Overall response rate is defined as response (CR, CRi or PR) at cycle 3 or cycle 6 evaluation. Only patients who completed at least 3 cycles were eligible for analysis for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oratumumab and Lenalidomide
Number analyzed (Participants) | 19
percentage of participants | 53 [32 to 73]

2. Secondary Outcome: Frequency of Adverse and Severe Adverse Events
Description: Frequency of adverse and severe adverse events
Time Frame: 30 weeks
Population: Adverse Events were assessed at each treatment visit. All patients who were treated are included in the adverse event analysis.
Measure: Number; unit: participants
Groups:
- Oratumumab and Lenalidomide: Single arm, non randomized study
  Ofatumumab, Lenalidomide: -Ofatumumab 2000 mg (300 mg on first cycle) IV on day 1.
  * Lenalidomide 10 mg (5 mg on first cycle) PO days 8-28.
  * Treatment to be administered for up to 6 cycles
  Ofatumumab: -Ofatumumab 2000 mg (300 mg on first cycle) IV on day 1 for up to 6 cycles (28 day cycles)
  -Treatment to be administered for up to 6 cycles
  Lenalidomide: -Lenalidomide 10 mg (5 mg on first cycle) PO days 8-28 for up to 6 cycles (28 day cycles)
Arm/Group | Oratumumab and Lenalidomide
Number analyzed (Participants) | 21
participants
  Number of SAEs | 4
  Neutropenia | 19
  grade 3/4 neutropenia | 10
  thrombocytopenia | 15
  grade 3/4 thrombocytopenia | 4
  tumor flare reaction | 9
  grade 3 tumor flare reaction | 1

3. Secondary Outcome: Biomarkers Changes During Treatment.
Description: Biomarkers changes during treatment. A minimum of 5 subjects will be enrolled in the biomarkers sub-study. Only those subjects enrolled at MUSC will be considered for the biomarkers sub-study. At day 1 of cycle 1, day 8 of cycle 1, day 1 of cycle 2 and day 8 of cycles 2, blood samples will be obtained for assessment of biomarkers.
Time Frame: 30 Weeks
Population: The biomarker sub-study was not completed due to poor accrual to this substudy and lack of feasibility.
Arm/Group | Oratumumab and Lenalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency of Adverse Events
Description: Number of adverse events occuring in greater than 20% of subjects
Time Frame: 30 weeks
Population: as for outcome 2
Measure: Number; unit: events
Arm/Group | Oratumumab and Lenalidomide
Number analyzed (Participants) | 21
events | 15

5. Secondary Outcome: Dose Reductions Due to Adverse Events.
Description: Number of dose reductions due to toxicity.
Time Frame: 30 weeks
Population: as for outcome 2
Measure: Number; unit: dose reductions
Arm/Group | Oratumumab and Lenalidomide
Number analyzed (Participants) | 21
dose reductions | 17

ADVERSE EVENTS:
Description: All subjects enrolled on study were evaluated for toxicity.
Arm/Group | Oratumumab and Lenalidomide
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oratumumab and Lenalidomide (N=21)
ALT Increase (Investigations) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oratumumab and Lenalidomide (N=21)
Neutrophil count decreased (Investigations) | 19
Platelet count decreased (Investigations) | 15
fatigue (General disorders) | 11
Tumor flare reaction (General disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
hypernatremia (Metabolism and nutrition disorders) | 8
Infusion related reaction (General disorders) | 7
dizziness (Nervous system disorders) | 7
hyperglycemia (Metabolism and nutrition disorders) | 7
Tachycardia (Cardiac disorders) | 7
Aspartate aminotransferase increased (Investigations) | 7
creatinine increased (Investigations) | 9
cough (Respiratory, thoracic and mediastinal disorders) | 6
hypoalbuminemia (Metabolism and nutrition disorders) | 7
lactic dehydrogenase increased (Investigations) | 6
Anemia (Blood and lymphatic system disorders) | 14
Night Sweats (General disorders) | 5
hypocalcemia (Metabolism and nutrition disorders) | 5
insomnia (Psychiatric disorders) | 4
nausea (Gastrointestinal disorders) | 4
fever (General disorders) | 4
Alanine amniotransferase increased (Investigations) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
pallor (General disorders) | 3
hypophosphatemia (Metabolism and nutrition disorders) | 3
constipation (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 3
leg cramps (Musculoskeletal and connective tissue disorders) | 4
diarrhea (Gastrointestinal disorders) | 3
Blood bilirubin increased (Investigations) | 3
hyperphosphatemia (Investigations) | 4
hypermagnesemia (Investigations) | 3
hyperuricemia (Metabolism and nutrition disorders) | 5
hypotension (Vascular disorders) | 3
weakness (Musculoskeletal and connective tissue disorders) | 3
alkaline phosphatase increased (Investigations) | 5
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
chills (General disorders) | 2
hypokalemia (Metabolism and nutrition disorders) | 2
Bradycardia (Cardiac disorders) | 2
anorexia (Metabolism and nutrition disorders) | 3
acute renal failure (Renal and urinary disorders) | 2
hypomagnesemia (Metabolism and nutrition disorders) | 2
wheezing (Respiratory, thoracic and mediastinal disorders) | 2
chloride increased (Metabolism and nutrition disorders) | 3
CO2 content decreased (Investigations) | 3
abdominal pain (Gastrointestinal disorders) | 2
non-cardiac chest pain (General disorders) | 1
actinic keratosis (Skin and subcutaneous tissue disorders) | 1
hypertension (Vascular disorders) | 4
hot flashes (Vascular disorders) | 2
back pain (Musculoskeletal and connective tissue disorders) | 3
uric acid decreased (Investigations) | 1
hypogammaglobulinemia (Investigations) | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 3
dysgeusia (Nervous system disorders) | 1
edema face (General disorders) | 1
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
pruritis (Skin and subcutaneous tissue disorders) | 1
irregular heartbeat (Cardiac disorders) | 1
lymphadenopathy (Infections and infestations) | 1
neck pain (Musculoskeletal and connective tissue disorders) | 1
lymph node pain (Immune system disorders) | 4
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
vomiting (Gastrointestinal disorders) | 1
white blood cell decreased (Investigations) | 1
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
weight loss (Investigations) | 1
alopecia (Skin and subcutaneous tissue disorders) | 1
bruising (Injury, poisoning and procedural complications) | 1
dry eye (Eye disorders) | 1
flushing (Vascular disorders) | 1
itchy eye (Eye disorders) | 1
pulmonari emboli (Vascular disorders) | 1
renal insufficiency (Renal and urinary disorders) | 1
watering eyes (Eye disorders) | 1
agitation (Psychiatric disorders) | 1
muscle cramping (Musculoskeletal and connective tissue disorders) | 2
espophagitis (Gastrointestinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 2
sinus tachycardia (Cardiac disorders) | 1
pneumonia (Infections and infestations) | 3
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 2
dry skin (Skin and subcutaneous tissue disorders) | 1
chloride decreased (Investigations) | 1
blood protein decreased (Investigations) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
sunburn (Skin and subcutaneous tissue disorders) | 1
sweating (General disorders) | 1
swollen feeling (General disorders) | 1
cellulitis (Infections and infestations) | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
mood swings (Psychiatric disorders) | 1
rash maculopapular (Skin and subcutaneous tissue disorders) | 1
rash (NOS) (Skin and subcutaneous tissue disorders) | 1
dehydration (Metabolism and nutrition disorders) | 1
hypercalcemia (Metabolism and nutrition disorders) | 1
paresthesia (Nervous system disorders) | 1
heartburn (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes